CLINICAL TRIAL: NCT02554266
Title: A Prospective, Multicenter, Single Arm Real-World Registry Investigating the Clinical Use and Safety of the Lutonix Drug Coated Balloon Percutaneous Transluminal Angioplasty (PTA) Catheter for Treatment of Below-the-Knee (BTK) Arteries
Brief Title: Registry Investigating the Clinical Use and Safety of the Lutonix Drug Coated Balloon for Treatment of BTK Arteries
Acronym: BTKRegistry
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0024-01
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Lutonix 014 Drug Coated Balloon PTA Catheter — Drug Coated Balloon PTA Catheter for Treatment of Below-the-Knee (BTK) Arteries

SUMMARY:
The study will enroll patients presenting with claudication, or critical limb ischemia (Rutherford Category 3- 5) and an angiographically significant (≥ 70%) native artery lesion appropriate for angioplasty that is below the knee. Subjects will be treated with the Lutonix Drug Coated Balloon (DCB) carrying the CE Mark per current IFU and followed clinically for a minimum of 2 years.

DETAILED DESCRIPTION:
Patients will be treated according to hospital routine with anticipated visits 30 days, 6 months, 12months and 24 months after the index procedure. Data on Rutherford grade, wound healing, patency of the target lesion, concomitant antiplatelet medication and Adverse Events will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breastfeeding female ≥18 years of age;
2. Rutherford Clinical Category 3-5;
3. Patient is willing to provide informed consent, and is willing to comply with the protocol-required follow up visits and recommended medication regimen;
4. Significant stenosis (≥70%) or occlusion of one or more native artery(s) below the tibial plateau and above the tibiotalar joint appropriate for angioplasty per operator visual assessment;
5. Lesion(s) can be treated with available Lutonix DCB device size matrix per current Instructions for Use (IFU); and
6. Target vessel(s) reconstitute(s) at or above the ankle with inline flow to at least one patent (<50% residual stenosis) inframalleolar outflow vessel (planned treatment below-the-ankle is not allowed).

NOTE: Outflow must be assessed AFTER pre-dilatation NOTE: More than one artery allowed, but each target vessel MUST demonstrate inline inframalleolar outflow.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Patient is currently participating in an investigational drug or device study which has not yet reached its primary endpoint or was previously enrolled into this registry (i.e. Lutonix BTK registry);
2. Inability to take recommended medications as stated in the IFU or non-controllable allergy to contrast; or
3. Neurotrophic ulcer or heel pressure ulcer or ulcer potentially involving calcaneus (index limb).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients presenting with claudication, or critical limb ischemia (Rutherford Category 3- 5) and an angiographically significant (≥ 70%) native artery lesion appropriate for angioplasty that is below the knee.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse limb related events below the knee and of perioperative death. | 30-days
  Freedom from the composite of all-cause death, above-ankle amputation or major reintervention, i.e. new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis, of the index limb involving a below-the-knee artery. All these events will be adjudicated by a Clinical Events Committee.
Rate of Target Lesion Revascularization (TLR) | 6 months
  Defined as clinically-driven target lesion reintervention. All re-interventions at the target limb are captured and adjudicated by a Clinical Events Committee.

SECONDARY OUTCOMES:
Primary patency of the target lesion | 6, 12 and 24 months
  Primary Patency of the target vessel is defined as freedom from total occlusion. Primary patency is assessed by the investigators.
Freedom from clinically-driven Target Lesion Revascularization (TLR) | 12 and 24 months
  All events leading to re-interventions at the target limb will be adjudicated by a Clinical Events Committee.
Rate of amputations above the ankle at the target limb | 1, 6, 12 and 24 months
  All events leading to amputations at the target limb will be adjudicated by a Clinical Events Committee.
Rate of Target vessel reintervention (TVR) | 1, 6, 12 and 24 months
  All events leading to re-interventions at the target limb will be adjudicated by a Clinical Events Committee.
Rate of unexpected device or drug-related adverse events | 1, 6, 12 and 24 months
  Unexpected device or drug-related adverse events are those events that are related to the device or drug, but are not listed in the potential adverse event section of the Instructions For Use.
Rate of reintervention for treatment of thrombosis of the target vessel(s) | 1, 6, 12 and 24 months
  Arteries may occlude from thrombosis
Rate of reintervention for embolization to its distal vasculature | 1, 6, 12 and 24 months
  Atherothrombotic debris may occlude the artery downstream and cause distal embolization.
Rate of death | 1, 6, 12 and 24 months
  All events leading to a patient's death will be adjudicated by a Clinical Events Committee.
Status of ischemic wounds at the target limb | 6 and 12 months
  Ischemic wounds and their status during the follow-up period will be captured.
Rate of new or recurrent artery lesions at the target limb | 6 and 12 months
  Artery lesions are captured as Adverse Events.
Change in Rutherford Class at the target limb | 6 and 12 months
  The Rutherford class is captured from Baseline to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Universitätsklinikum Leipzig: Angiologie; Michael Lichtenberg, MD, Principal Investigator — Klinikum Arnsberg
Locations (26):
- Austria (4):
  - LKH-Univ. Klinikum Graz, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medical University Vienna, Department of Angiology, Vienna
  - Medical University Vienna, Department of Radiodiagnostic, Vienna
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - AZ Groeninghe, Kortrijk
- Hôpital européen Georges-Pompidou, Paris, France
- Germany (8):
  - Klinikum Hochsauerland, Arnsberg
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Rechts der Isar, Munich
  - Marienhospital Osnabrück, Osnabrück
  - Klinikum Rosenheim, Rosenheim
  - MEDINOS Klinik Sonneberg, Sonneberg
  - Kreiskrankenhaus Viechtach, Viechtach
- Greece (2):
  - Attikon University Hospital, Athens
  - Patras University Hospital, Pátrai
- Italy (3):
  - Clinica Montevergine, Mercogliano
  - Policlinico di Monza, Monza
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- Hospital Santa Marta (C.H.Lisboa Central), Lisbon, Portugal
- King Faisal Hospital and Medical research Center, Riyadh, Saudi Arabia
- Corporación Sanitaria Parc Taulí, Sabadell, Spain
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zurich, Zurich
- University Hospital of South Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No